CLINICAL TRIAL: NCT01086566
Title: Evaluation of the Safety and Cellular and Humoral Immune Response to Primary and Secondary Immunization With Subvirion H5N1 Vaccines Representing Different Clades
Brief Title: Cellular and Humoral Immune Response to Primary and Secondary Immunization With Subvirion H5N1 Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 08-0059; UR revax CMI
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: Influenza, H5N1, avian influenza, parent protocol
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (5):
- Multiple Boost Group-15 mcg (Experimental): 25 healthy adults who have previously received both Clade 1 and Clade 3 vaccines as a participant in study DMID 05-0043 will receive a single dose of 15 mcg of A/Indonesia/5/05.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005
- Primed Group-15 mcg (Experimental): 30 healthy adults who have previously received H5N1 vaccine at any dose will receive a single dose of 15 mcg of A/Indonesia/5/05.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005
- Unprimed Group-90 mcg (Experimental): 15 healthy adults with no previous receipt of H5N1 vaccine at any dose will receive 2 doses of 90 mcg of A/Indonesia/5/05 vaccine separated by 28 days.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005
- Unprimed Group-15 mcg (Experimental): 15 healthy adults with no previous receipt of H5N1 vaccine at any dose will receive 2 doses of 15 mcg of A/Indonesia/5/05 vaccine separated by 28 days.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005
- Primed Group-90 mcg (Experimental): 30 healthy adults who have previously received H5N1 vaccine at any dose will receive a single dose of 90 mcg of A/Indonesia/5/05.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005

INTERVENTIONS:
Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Indonesia/05/2005 — Inactivated monovalent subvirion H5N1 vaccine (HA of A/Indonesia/05/05) provided in unit-dose vials containing 0.5 mL of either 30 mcg/mL A/H5N1 HA or 180 mcg/mL A/H5N1 HA. Subjects will receive 1 of 2 dose levels of vaccine, 15 or 90 mcg.

SUMMARY:
The purpose of the study is to evaluate safety and compare how the body reacts to 2 different strengths of the Clade (specific type of H5N1 virus) 2 H5N1 flu vaccine when given as a single vaccination with a high dose (90 mcg) or low dose (15 mcg) to volunteers who have received at least 2 doses of the Clade 1 H5N1 vaccine, in a previous National Institute of Health study or who have never received a H5N1 vaccine (naïve). Previously vaccinated subjects (in studies 04-0063, 05-0090, 05-0127) will receive either 15 or 90 mcg of H5N1 vaccine. Multiply boosted volunteers who participated study 05-0043 and received Clade 1 and 3 vaccines, will receive the same dose (15mcg). Vaccine naïve subjects will receive 2 doses of vaccine (15 or 90 mcg) separated by 28 days. Blood samples will be collected. 115 volunteers age 18-64 may participate in study related procedures for approximately 7 months.

DETAILED DESCRIPTION:
In response to the steadily increasing number of reports of human infection with avian influenza A (H5N1) viruses, there is now a world-wide effort to develop and test potential candidate vaccines for this and other avian viruses with pandemic potential. The study will be conducted as a laboratory blinded assessment of the humoral and cellular immune response to A/Indonesia/5/05 vaccine in three populations: healthy adults who have previously received a clade 1 H5 vaccine in a Division of Microbiology and Infectious Diseases (DMID)-sponsored study; healthy adult recipients of prime-boost regimens representing two clades; and healthy adults with no previous H5 vaccination and who are not at risk for H5 exposures. Primed subjects are randomized to receive a single dose of either 15 mcg or 90 mcg of A/Indonesia/5/05 vaccine. Multiply boosted subjects are those who participated in study 05-0043, and have previously received both A/HK/97 (Clade 3) and A/VN/04 (Clade 1) vaccines. Because only a small number of such subjects are available, they will not be randomized but will all receive the same dose of vaccine. Unprimed subjects are randomized to receive 2 doses of 15 mcg or 90 mcg of A/Indonesia/5/05 vaccine separated by 28 days. In all groups, sera and peripheral blood mononuclear cells (PBMC) are obtained prior to and on days 3, 7, 14, and 28 after each dose. Primed and multiply boosted subjects also have sera and PBMC obtained on day 56. All groups will make a final study visit at 6 months following the last dose of vaccine (day 180 for primed and boosted subjects and day 208 for unprimed subjects). Approximately 115 subjects between the ages of 18 and 64 will participate in this study. The primary objective is to determine the safety of administration of the A/Indonesia/05 subvirion vaccine when administered to healthy, primed or unprimed adults. The secondary objective is to: determine the effects of priming with a clade 1 vaccine on antibody responses to revaccination with a clade 2 vaccine. The tertiary objectives are to determine the effects of priming on the repertoire and phenotypes of B and T cells generated in response to vaccination; to evaluate whether pre-existing immunity to seasonal influenza viruses impacts the specificity and magnitude of the cluster of differentiation marker (CD)4 T cell response to H5 vaccination and to describe the kinetics of the cellualr immune response to subvirion H5N1 vaccinatin in primed and unprimed individuals. The primary endpoint is reactogenicity, adverse event (AE) and serious adverse event (SAE) information, solicited in-clinic and via memory aids. The secondary endpoints are: levels of HAI antibody recognizing A/Indonesia/05 (Clade 2), A/Vietnam/04 (Clade 1) and representative Clade 2 subclade viruses, and levels of neutralizing antibody assessed by neutralization tests using the rgA/Indonesia/5/05 virus prior to and Days 3, 7, 14, and 28 after each vaccination. This study is linked to DMID protocols 04-063, 05-0090, 05-0043 and 05-0127.

ELIGIBILITY:
Inclusion Criteria:

* To participate in the primed group, the subject must have previously received at least 2 doses via the intramuscular route of subvirion inactivated A/H5N1/VN/1203/04 (H5N1) vaccine as part of a Division of Microbiology and Infectious Diseases (DMID)-sponsored protocol.
* To participate in the multiple boost group, the subjects must have previously received both clade 1 and clade 3 vaccines as a participant in the DMID 05-0043 study.
* To participate in the unprimed group, the subject must not have received previous H5N1 vaccine at any dose.
* The subject must be between the ages of 18 and 64 years, inclusive.
* Female subjects must fulfill one of the following: (i) not able to bear children because she has been surgically sterilized (tubal ligation or hysterectomy) for at least one year or is at least 1 year post-menopausal or (ii) agrees to practice effective methods of contraception that may include, but are not limited to abstinence, barrier methods, monogamous relationship with vasectomized partner, birth control pills, patches, hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices), from 30 days prior to study enrollment through 30 days following receipt of the last dose of vaccine.
* Female subjects of childbearing potential must have a negative pregnancy test (urine or serum) within 24 hours prior each to vaccination.
* The subject must be in good health, as determined by: vital signs (heart rate <100 beats per minute (bpm); blood pressure: systolic greater than or equal to 90 mm Hg and less than or equal to 140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature <100.0 degrees Fahrenheit); medical history; and targeted physical examination, when necessary, based on medical history. Stable medical condition is defined as: no recent change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc, or is done for financial reasons, as long as in the same class of medication, will not be considered a violation of the inclusion criterion. Any change to prescription medication due to improvement of a disease outcome will not be considered a violation of the inclusion criterion.
* The subject is able to understand and comply with the planned study procedures, including being available for all study visits.
* The subject has provided informed consent prior to any study procedures.

Exclusion Criteria:

* The subject is allergic to eggs, egg products, chicken or egg proteins or other components of the vaccine (including gelatin, formaldehyde, octoxinol and thimerosal).
* The subject is a woman who is breastfeeding or intends to become pregnant during the study period between enrollment and 30 days following receipt of the last dose of vaccine.
* The subject is immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* The subject has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy. For this criterion, "active" is defined as having received treatment within the past 5 years.
* The subject has long-term (> 2 weeks) use of oral or parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* The subject received immunoglobulin or another blood product within the 3 months prior to enrollment in this study.
* The subject has received an inactivated vaccine within the 2 weeks or a live vaccine within the 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days (or 56 days for vaccine naïve recipients).
* The subject has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include, but are not limited to: solicited reactogenicity symptoms, history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); subjects with diabetes mellitus, well-controlled with oral agents may enroll as long as there has been no dose adjustment with the past 6 months; insulin-dependent diabetes is excluded; cardiac insufficiency, if heart failure is present (New York Association Functional Class III or IV); an atherosclerotic event during the 6 months prior to enrollment (e.g., history of myocardial infarction, stroke, recanalization of femoral arteries or transient ischemic attack).
* The subject has a history of a severe reaction following receipt of an influenza virus vaccine.
* The subject has an acute illness or an oral temperature greater than 99.9 °F (37.7 °C) within 3 days prior to enrollment or vaccination. Subjects who had an acute illness that was treated symptoms resolved are eligible to enroll as long as treatment is completed and symptoms resolve > 3 days prior to enrollment.
* The subject is currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study, or intends to donate blood during the study period.
* The subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* The subject has a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis.
* The subject has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* The subject is receiving psychiatric drugs. Psychiatric drugs include, but are not limited to: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensation are allowed enrollment into the study.
* The subject has a history of alcohol or drug abuse in the 5 years prior to enrollment.
* The subject has a known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* The subject has a history of Guillain-Barré syndrome.
* The subject has any condition that the investigator believes may interfere with successful completion of the study.
* The subject has occupational exposure to live H5N1 viruses or has received an H5N1 vaccine outside of the context of a DMID study. Subjects with a previous history of receipt of an H5N1 vaccine in an oil-in-water emulsion adjuvant are also excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reactogenicity: Occurrence of vaccine-associated unsolicited adverse events through Day 28 after the last vaccination | Day 0 to Day 28 for primed and boosted subjects and Day 0 to Day 56 for unprimed subjects.
Reactogenicity: Occurrence of vaccine-associated solicited local and systemic adverse events within 8 days post-vaccination (Day 0-7) | Within 8 days post-vaccination (Day 0-7)
Reactogenicity: Occurrence of vaccine-associated unsolicited serious adverse events (SAEs) through the course of the study | Day 0 through 6 months after last dose of vaccine (day 180 for primed and boosted subjects and day 208 for non-primed subjects)

SECONDARY OUTCOMES:
Levels of HAI antibody recognizing A/Indonesia/05 (Clade 2), A/Vietnam/04 (Clade 1) and representative Clade 2 subclade viruses prior to and Days 3, 7, 14, and 28 after each vaccination in primed and unprimed subjects. | Blood samples taken prior to vaccination on Day 0, and approximately 3, 7, 14, and 28 days after each dose of vaccine in primed and unprimed subjects
Levels of neutralizing antibody assessed by neutralization tests using the rgA/Indonesia/5/05 virus prior to and Days 3, 7, 14, and 28 after each vaccination. | Blood samples taken prior to vaccination on Day 0, and approximately 3, 7, 14, and 28 days after each dose of vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York, United States